CLINICAL TRIAL: NCT04027907
Title: Platelet Activity in Type 2 Diabetic Patients Using Flowcytometry in Relation to Macrovascular Complication.
Brief Title: Platelet Activity in T2DM Using Flowcytometry
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hanaa M Ahmed, HMAmed, Assiut University
Other Study IDs: Plt activity by flowcytometry
Record Dates: First submitted 2019-07-18; First posted 2019-07-22 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Platelet Activity in T2DM Using Flowcytometry

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- T2DM
  Interventions: Other: Flowcytometry
- healthy controls
  Interventions: Other: Flowcytometry

INTERVENTIONS:
Other: Flowcytometry — detect platelet activity in T2DM by surface expression of platelet receptors determined by flowcytometry using different monoclonal antibodies (CD62 and CD63).

SUMMARY:
-Describe platelet activity in type 2 diabetes as a participant in vascular inflammation. -Compare platelet activity in patients with type 2 diabetes mellitus versus healthy controls. -Study and describe platelet activity in patients with type 2 diabetes mellitus in association with ischemic cardiovascular disease in relation to duration of diabetes mellitus .

DETAILED DESCRIPTION:
Type2diabetes mellitus(T2DM)is most prevalent and costly chronic disease(Leon et al 2015).according to IDF a further increase to 642million diagnosed individual by2040(Ogurtsova et al 2017).the major cause of morbidity and mortality in DM is macrovascular complications.75% of diabetic patients die of cardiovascular disease(CVD)( Ridker et al2017).Platelets are one of blood cells 1,5-3um in size and survive 8-10days ,their function extended beyond homestasis and thrombosis to be an active participant in intiating and sustaining vascular inflammation as well as in prothrombotic complications of CVD(Festa et al2002).platelets are hyperactive in diabetic patients ,the coagulation cascade is dysfunctional ,platelet inT2DM adhere to vascular endothelium and aggregate more readily than those in healthy people(Pretorius2011)*.platelets are activated when they are in contact with damaged vascular endothelium , once activated they secrete awide spectrum of inflammatory mediators , once they are activated , they intiate reactions by changes in the level of expression of surface glycoproteins(GP)results , which act as receptors for platelet agonist and for adhesive proteins involved in platelet aggregation(Pretorius etal2015)**.platelet activity can be measured by flow cytometry ,as flow cytometry allows the simultaneous detection of surface antigens in a sensitive and specific manner , it is therefore possible to examine aspects of the platelet membrane activity . the available platelet markers areCD41a marker forGP2b ,CD42 a marker for GP1b.both are used for platelet identification.( Pretorius et al 2017)***.CD62 a marker for P-selectin ,anti-CD62 react with alpha granule membrane protein which is expressed on the surface of activated platelet.CD63 a marker for GP4 and anti-CD63 react with lysosomal granule-membrane glycoprotein that is expressed on surface of activated platelet. CD62andCD63 are markers of platelet activation (Ibrahim et al 2017).knowing the major role of platelets in inflammatory and healing process in the vascular system especially in diabetic patients ,created the urgency to study the impact of platelet activity in diabetic patients whom has macrovascular risk using flowcytometry.

ELIGIBILITY:
Inclusion Criteria:

* The study will include patient with type II diabetes at age of 30-60 years old with or without ischemic cardiovascular disease. . Controls will be healthy individuals with normal blood glucose level of same matched age group.

Exclusion Criteria: 1)Type1Diabetes mellitus. 2)Hypertensive patients. 3)patients with renal impairment. 4) patients with hepatic impairment. 5)patients with thrombocytopenia. 6)Pregnancy.

Ages: 30 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Diabetic patients will be recruited from Internal medicine department and Diabetes out patient clinic in Assuit University Hospital.
  Controls will be health workers and paramedicals in Assuit university hospital.
Sampling Method: Non-Probability Sample
Enrollment: 122 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Platelet activity in type 2 diabetic patients using flowcytometry in relation to macrovascular complication. | Baseline
  Dedect platelet activity by surface expression of platelet receptors determined by flowcytometry using different monoclonal antibodies (CD62 and CD63)

SECONDARY OUTCOMES:
Platelet activity in type 2 diabetic patients using flowcytometry in relation to macrovascular complication. | Baseline
  Dedect platelet number by surface expression of platelet receptors determined by flowcytometry using different monoclonal antibodies (CD41 and CD42)

CONTACTS AND LOCATIONS:
Overall Officials: hanaa ahmed, master, Principal Investigator — Assiut University

REFERENCES:
- [Result] Castaigne F, Liber E, Carbillet L, Boulet M, Riel RR. [New procedure for protein spinning: the hydrodynamic process]. Ann Nutr Aliment. 1978;32(2-3):217-31. French. PMID 707914
- [Result] Gulati RB, Wadia RS, Shaikh RA, Soares PM, Grant KB. Precordial mapping in acute myocardial infarction. Jpn Heart J. 1977 Jul;18(4):447-56. doi: 10.1536/ihj.18.447. PMID 909154
- [Result] Gheorghiu T, Badescu A. [Dynamcis of immunocompetent cells in the contralateral lymph node in grafted cancer, under the influence of some factors stimulating and inhibiting the CNS in rats]. Rev Med Chir Soc Med Nat Iasi. 1976 Jan-Mar;80(1):79-84. No abstract available. Romanian. PMID 9680